CLINICAL TRIAL: NCT02009982
Title: Cardioneuroablation for Neurocardiogenic Syncope
Acronym: Ablate-NCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David B. De Lurgio (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor-Investigator, David B. De Lurgio, Associate Professor of Medicine, Emory University
Organization: Emory University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00062061
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Results first posted 2016-11-04 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-09

CONDITIONS: Neurocardiogenic Syncope; Vasovagal Syncope
Keywords: Fainting; Ablation; Cardiology; Cardiac Electrophysiology
MeSH Terms: conditions — Syncope, Vasovagal; Syncope

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cardioneuroablation (Experimental): Patients in this group will receive the cardioneuroablation procedure using the Biosense Webster Navistar ThermoCool Diagnostic/Ablation Deflectable Tip Catheter
  Interventions: Procedure: Cardioneuroablation; Device: Biosense Webster Navistar ThermoCool Diagnostic/Ablation Deflectable Tip Catheter
- Standard Medical Thearpy (No Intervention): Patients in this group will not receive the cardioneuroablation and will continue to be managed using standard medical therapy

INTERVENTIONS:
Procedure: Cardioneuroablation — Catheter Ablation of Vagal Inputs in Left Atrium
  Arms: Cardioneuroablation
Device: Biosense Webster Navistar ThermoCool Diagnostic/Ablation Deflectable Tip Catheter — This is the device that will be used to perform the Cardioneuroablation procedure
  Arms: Cardioneuroablation

SUMMARY:
The purpose of this study is to evaluate the effectiveness of cardioneuroablation for the treatment of neurocardiogenic syncope (NCS), also known as "vaso-vagal" syncope. Syncope is a general term for passing out spells and neurocardiogenic syncope is a specific form of passing out spells caused by sudden drops in heart rate or blood pressure. Although the specific mechanisms of NCS are not well understood, it is believed that some people are prone to developing passing out spells in specific situations such as standing up for a long period of time, pain or nausea. In these situations, the body reacts with a paradoxical reflex which leads to a drop in blood pressure and heart rate and causes passing out. Certain types of medications are used to treat NCS including beta-blockers, midodrine and florinef, among others. However, none of these medications are particularly effective at preventing passing out spells and many people continue to have episodes despite trying different medications.

Cardioneuroablation is a new form of treatment for NCS. The term ablation means using a wire to make small electrical burns in the heart. Ablation has been used for many years to treat other electrical disturbances in the heart but the use of ablation to treat NCS is a new application. The goal of cardioneuroablation is to identify areas within the heart which are believed to initiate the reflex which triggers the drop in heart rate and blood pressure that leads to passing out. In preliminary studies, it has been suggested that cardioneuroablation may be significantly more effective than medications at preventing passing out spells for people with NCS.

Hypothesis: Cardioneuroablation of vagal inputs in the left atrium may serve as an effective treatment modality for the prevention of NCS by blunting the initial trigger of the cascade that leads to symptoms and syncope.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able and willing to sign and date the Patient Consent Form
* Subject is 18 years of age or older
* Subject is expected to remain available for the follow-up protocol
* Subject is willing to comply with the follow-up procedures
* Subject has medically documented history of neurocardiogenic syncope
* Subject has had 3 episodes of syncope or presyncope in last 12 months
* Subject has had a positive tilt table test, defined as the presence of syncope or presyncope associated with abrupt hypotension (SBP < 70 mmHg) or bradycardia (HR < 40 bpm), with or without sublingual nitroglycerin provocation or atropine challenge
* Subject has been tried on at least one pharmacologic therapy for at least 4 weeks

Exclusion Criteria:

* Subject has signs and symptoms of an active infection (i.e. fever, elevated white blood cell count, etc.) which has not been treated and/or has not demonstrated improvement in white blood cell count and resolution of fever
* Subject is pregnant or planning to become pregnant within the study protocol follow-up
* Subject is enrolled or planning to participate in a concurrent drug and/or device study during the course of this study that would confound study results as determined by the study physician
* Subject is unwillingly to comply with the randomization procedure
* Subject has had no syncopal episodes in last six months while on medical therapy
* Subject has one of the following conditions that is the documented source of syncope: sick sinus syndrome, sinus node or atrioventricular conduction deficiencies, ventricular tachyarrhythmias, pulmonary hypertension, hypertrophic cardiomyopathy, history of transient ischemic attack, seizure disorders, subclavian steal syndrome, or drug-induced syncope
* Subjects with a myocardial infarction within last six months
* Subjects with severe heart failure (NYHA class III or IV), previous heart surgery, structural heart disease, or an infiltrative cardiac disease
* Subject is contraindicated for left-atrial ablation, as determined by enrolling physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David B DeLurgio, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University, Atlanta, Georgia
  - University of North Carolina, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No
No due to limited data set and study ending.

RESULTS

PARTICIPANT FLOW:
Groups:
- Cardioneuroablation: Patients in this group received the cardioneuroablation procedure using the Biosense Webster Navistar ThermoCool Diagnostic/Ablation Deflectable Tip Catheter
  Cardioneuroablation: Catheter Ablation of Vagal Inputs in Left Atrium
  Biosense Webster Navistar ThermoCool Diagnostic/Ablation Deflectable Tip Catheter: This is the device that was used to perform the Cardioneuroablation procedure
- Standard Medical Thearpy: Patients in this group did not receive the cardioneuroablation and were managed using standard medical therapy.
Period: Overall Study
Arm/Group | Cardioneuroablation | Standard Medical Thearpy
Started | 1 | 2
Completed | 1 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cardioneuroablation | Standard Medical Thearpy | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 3
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Syncope Recurrence Rate
Description: The primary endpoint for the study is recurrence of syncope within the 12 month follow-up protocol
Time Frame: 12 Months
Population: No data was analyzed due to low enrollment.
Arm/Group | Cardioneuroablation | Standard Medical Thearpy
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Incidence of Serious Adverse Events
Description: The secondary endpoint for this study will be the incidence of serious adverse events related to the study procedure within the 12 month follow-up protocol
Time Frame: 12 Months
Population: No data was analyzed due to low enrollment.
Arm/Group | Cardioneuroablation | Standard Medical Thearpy
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Data for adverse events were collected for 12 months.
Arm/Group | Cardioneuroablation | Standard Medical Thearpy
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 1/1 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cardioneuroablation (N=1) | Standard Medical Thearpy (N=2)
Chest Pain (Cardiac disorders) | 1 (1) | 0 (0)
Tremors (Nervous system disorders) | 1 (1) | 0 (0)
Upper Respiratory Infection (Infections and infestations) | 1 (2) | 0 (0)
Angina (Cardiac disorders) | 1 (1) | 0 (0)
Edema (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Shingles (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes